CLINICAL TRIAL: NCT02446860
Title: A Study of Anti-PD1 (Nivolumab) Therapy as Pre- and Post-operative Therapy in Metastatic Renal Cell Cancer (ADAPTeR)
Acronym: ADAPTeR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was unable to recruit the target number of patients (enrolled 15 instead of 19) and did not extend recruitment.
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CCR 4151
Record Dates: First submitted 2015-03-12; First posted 2015-05-18 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nivolumab (Experimental): Nivolumab 3 mg/kg by intravenous infusion, given every two weeks for eight weeks prior to nephrectomy, then post-operatively until patient is no longer deriving clinical benefit
  Interventions: Drug: nivolumab

INTERVENTIONS:
Drug: nivolumab — Nivolumab 3 mg/kg by intravenous infusion, given every two weeks for eight weeks prior to nephrectomy, then post-operatively until patient is no longer deriving clinical benefit.
  Other Names: Opdivo

SUMMARY:
Single arm, open label, phase II trial. Participants to undergo biopsy of primary tumour followed by 8 weeks of nivolumab therapy followed by nephrectomy. Nivolumab to be continued post-operatively

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is diagnosed in around 8500 patients annually in the UK. Approximately one third of these patients present with metastatic disease where the RCC has spread to other organs. The mainstay of treatment for these patients is systemic drug therapy, but surgery to remove the primary kidney tumour (i.e. nephrectomy) may also provide clinical benefit.

There is no standard preoperative systemic drug therapy in metastatic RCC, but such preoperative therapy is used widely in the treatment of other cancer types. This approach has several potential advantages including shrinking the tumour to help improve surgical outcomes and to aid identification of appropriate postoperative Drug therapy.

Over the last 10 years several agents have demonstrated promising activity in RCC including the monoclonal antibody therapy nivolumab. This novel immunotherapy works by blocking an immune cell receptor (programmed death1(PD1)) which the cancer can otherwise utilise to evade an individuals immune system attack. This study will investigate the use of nivolumab therapy as a preoperative treatment in patients with metastatic RCC for whom nephrectomy is planned. A total of 19 patients will be recruited at the Royal Marsden Hospital Patients will be treated with nivolumab for 8 weeks prior to surgery, after which nivolumab therapy will restart and continue until such time that the patient is not receiving an overall clinical benefit.

The primary aim of the study will be to assess the safety of such a strategy, with further aims to assess clinical effectiveness. This is also a unique opportunity to further investigate the way in which nivolumab works and to identify predictors of treatment response. To achieve this patients will be asked to provide biopsy samples of their RCC pre & post nivolumab treatment and their nephrectomy tissue for research use, alongside additional blood & urine samples.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic renal cell carcinoma of predominately clear cell type
2. At least one site of disease outside the kidney measurable per RECIST 1.1
3. Scheduled to undergo nephrectomy as part of treatment plan
4. No prior systemic therapy for renal cell carcinoma
5. Male or female, 18 years of age or older
6. Life expectancy of 12 weeks or greater
7. ECOG performance status 0 or 1
8. Immunosuppressive doses of systemic medications, such as steroids or absorbed topical steroids (equivalent to 10 mg of prednisone daily or more) must be discontinued at least two weeks prior to administration of the study drug. Inhaled corticosteroids and adrenal replacement steroid doses of > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
9. Serum aspartate transaminase (AST) / serum alanine transaminase (ALT) ≤3x upper limit of normal (ULN)
10. Total serum bilirubin ≤1.5 x ULN (except subjects with Gilbert syndrome, who can have total bilirubin <3mg/dL (50µmol/L)
11. Serum creatinine ≤1.5 x ULN or creatinine clearance ≥40ml/min (measured or calculated using Cockcroft-Gault formula)
12. White blood cells (WBC) ≥ 2.0x109/L, Absolute neutrophil count (ANC) ≥1.5x109/L
13. Platelets ≥100 x109/L,
14. Haemoglobin ≥9.0 g/dL
15. Prothrombin time (PT) ≤1.5 x ULN
16. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment
17. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

1. Intracranial disease, unless there has been radiological evidence of stable intracranial disease > 6 months.
2. Need for nephrectomy to relieve symptoms relating to the primary tumour or for emergency nephrectomy
3. History of severe hypersensitivity reaction to other monoclonal antibodies
4. Prior malignancy, active within the last 3 years, except for locally curable cancers which have been apparently cured
5. Known HIV or AIDS-related illness
6. Any active, known or suspected autoimmune disease or any condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and physiological replacement doses >10mg daily prednisolone equivalent are permitted in the absence of active autoimmune disease.
7. Active infection requiring therapy
8. Positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA) indicating acute or chronic infection
9. Pregnancy or breastfeeding. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy and for 26 weeks following the last dose of study drug. All female patients with childbearing potential must have a negative pregnancy test (serum or urine) prior to enrolment/nivolumab treatment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy and for 31 weeks after the last dose of study drug. Women who are not of childbearing potential and azoospermic men do not require contraception.
10. Current signs or symptoms of severe progressive or uncontrolled hepatic, haematologic, gastrointestinal, endocrine, pulmonary or cardiac disease other than directly related to RCC
11. Use of vaccines against infectious diseases (eg influenza, varicella) within 28 days of initiation of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Safety profile of Nivolumab given pre- and post-nephrectomy in metastatic renal cell carcinoma. Safety will be assessed by a summary of adverse events and by the proportion of patients experiencing all grades of toxicity. | Until disease progression, measured every 2 weeks, on average for 11 months

SECONDARY OUTCOMES:
Response rate | Until progression or withdrawal of consent, measured every 8 weeks in first year and then every 12 weeks there after, on average for 11 months

OTHER OUTCOMES:
Progression free survival | Until progression or withdrawal of consent, measured every 8 weeks in first year and then every 12 weeks there after, on average for 11 months
Overall survival | Until death or withdrawal of consent, measured every 12 weeks, on average for 12 months
Changes in biomarkers | Until progression or withdrawal of consent, at cycle 1, pre-nephrectomy and at disease progression, on average for 11 months
  Changes in biomarkers correlated with both response to treatment and toxicity. This study aims to investigate the relation of ITH and the immune response to RCC in the context of PD-1 checkpoint-blockade, and to correlate putative immune biomarkers with clinical response or resistance in the pre-operative clinical trial 'window' model that has already been established.

CONTACTS AND LOCATIONS:
Overall Officials: James Larkin, Study Director — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The trial terminated early due to low recruitment and the small sample size 15 participants determined as insufficient for meaningful secondary analysis.

REFERENCES:
- [Background] Au L, Hatipoglu E, Robert de Massy M, Litchfield K, Beattie G, Rowan A, Schnidrig D, Thompson R, Byrne F, Horswell S, Fotiadis N, Hazell S, Nicol D, Shepherd STC, Fendler A, Mason R, Del Rosario L, Edmonds K, Lingard K, Sarker S, Mangwende M, Carlyle E, Attig J, Joshi K, Uddin I, Becker PD, Sunderland MW, Akarca A, Puccio I, Yang WW, Lund T, Dhillon K, Vasquez MD, Ghorani E, Xu H, Spencer C, Lopez JI, Green A, Mahadeva U, Borg E, Mitchison M, Moore DA, Proctor I, Falzon M, Pickering L, Furness AJS, Reading JL, Salgado R, Marafioti T, Jamal-Hanjani M; PEACE Consortium; Kassiotis G, Chain B, Larkin J, Swanton C, Quezada SA, Turajlic S; TRACERx Renal Consortium. Determinants of anti-PD-1 response and resistance in clear cell renal cell carcinoma. Cancer Cell. 2021 Nov 8;39(11):1497-1518.e11. doi: 10.1016/j.ccell.2021.10.001. Epub 2021 Oct 28. PMID 34715028